CLINICAL TRIAL: NCT03398434
Title: A Multicenter, Randomized, Open-label, Active-controlled, Dose-range Finding Study to Assess the Pharmacodynamic Parameters, Safety and Tolerability of MAA868 and Its Effect on Thrombogenesis Biomarkers Compared to Apixaban in Patients With Atrial Fibrillation
Brief Title: Efficacy and Safety of MAA868 in Patients With Atrial Fibrillation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial cancelled before First Patient First Visit (no patient enrolled)
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CMAA868A2202; 2017-002741-29 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
Keywords: MAA868; apixaban; atrial fibrillation; anticoagulant; Factor XI; D-dimer; systemic thromboembolic events
MeSH Terms: conditions — Atrial Fibrillation | interventions — MAA868; apixaban

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, blinded endpoint evaluation, active controlled, dose-range finding study.
Who Masked: Outcomes Assessor
Masking Description: blinded (with majuscule) endpoint evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MAA868 low dose regimen (Experimental): patients receive dose monthly.
  Interventions: Drug: MAA868
- MAA868 middle dose regimen (Experimental): patients receive dose monthly.
  Interventions: Drug: MAA868
- MAA868 high dose regimen (Experimental): patients receive dose monthly.
  Interventions: Drug: MAA868
- Apixaban (Active Comparator): Apixaban 5 mg b.i.d
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: MAA868 — 3 MAA868 doses, single administration, subcutaneous,
  Arms: MAA868 high dose regimen; MAA868 low dose regimen; MAA868 middle dose regimen
Drug: Apixaban — Apixaban 5 mg b.i.d
  Arms: Apixaban

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, pharmacodynamics, safety and tolerability of MAA868 compared to apixaban in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 55 and < 85 years old
* Body weight between 50 and 130 kg inclusive
* Atrial fibrillation or atrial flutter, as documented by electrocardiography
* CHA2DS2-VASc risk score ≥ 2 for male and female patients. Male patients with CHA2DS2VASc risk score of 1 can be included if anticoagulation therapy is warranted.
* Either anticoagulant-naïve or receiving a stable treatment of a recommended dose of a new oral anticoagulant (NOAC) over the 8 weeks prior to screening.

Exclusion Criteria:

* History of stroke, transient ischemic attack or systemic embolism
* History of major bleeding during treatment with an anticoagulant or antiplatelet therapy in the last 12 months
* History of traumatic or non-traumatic intracranial, intraspinal or intra-ocular bleeding
* Known bleeding diathesis or any known active bleeding site at screening or baseline
* Family history of bleeding disorder
* Known active GI lesions predisposing to bleeding events
* Myocardial infarction, unstable angina pectoris or coronary artery bypass graft (CABG) surgery within 12 months prior to the screening period
* Known hemodynamically significant valvular heart disease
* Uncontrolled hypertension defined as SBP/DBP ≥ 160/100 mmHg at the screening visit
* Heart failure NYHA class IV in the 3 months prior to the screening visit
* Dual antiplatelet therapy. Treatment with a P2Y12 inhibitor or low dose aspirin (≤ 100 mg/d) is allowed but not both.
* Severe renal impairment (creatinine clearance < 30 mL/min) at the screening visit

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-16 (Estimated); Primary Completion 2019-11-28 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
number of patients achieving FXI inhibition ≥ 80% at trough after monthly dosing at 3 dose levels of MAA868 inhibition | month 3
  Occurrence of achieving ≥ 80% inhibition of FXI (< 20% free FXI) following 3 months of treatment.

SECONDARY OUTCOMES:
number of patients achieving FXI inhibition ≥ 80% at trough after the first and second dose at 3 dose levels of MAA868 | Month 1 and 2
  Occurrence of achieving ≥ 80% inhibition of FXI (< 20% free FXI) at trough on Month 1 and Month 2
Number of patients with incidence of major or clinically relevant non-major (CRNM) bleeding events during the treatment period. | day 1 to day 91
  Incidence of major or clinically relevant non-major bleeding events
the effect of MAA868 on D dimer and other thrombogenesis biomarkers as indicators of efficacy compared to compotator | Days 31, 61 and 91
  Change from baseline to Day 31, Day 61 and Day 91 in thrombogenesis biomarkers (D-dimer, prothrombin fragment 1.2 (F1.2), thrombin-antithrombin III-complexes (TAT), fibrinogen).

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.